CLINICAL TRIAL: NCT07260591
Title: A Single-Arm, Open-Label, Compassionate Use Study of VSV-02 Administered Intravenously and Intratumorally in Patients With Advanced Solid Tumors
Brief Title: VSV-02 Compassionate Use in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSV-02A01tqyy
Record Dates: First submitted 2025-09-26; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Melanoma; Breast Cancer; Lung Cancer; Cancer Treatment; Immunotherapy
MeSH Terms: conditions — Melanoma; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VSV-02 Dose Escalation Group (Experimental): Participants will receive VSV-02 via intravenous (IV) and intratumoral (IT) injection in a dose-escalation manner. The starting dose is 6×10^10 PFU (IT) + 6×10^11 PFU (IV). Dosing occurs on Day 1 of each 21-day cycle for up to 6 cycles.
  Interventions: Biological: VSV-02 Injection

INTERVENTIONS:
Biological: VSV-02 Injection — VSV-02 Injection is an oncolytic virus vaccine based on an attenuated Vesicular Stomatitis Virus (VSV) that is engineered to encode a CD3/PD-L1 bispecific antibody. It is supplied as a sterile solution by Shanghai Rongrui Pharmaceutical Technology Co., Ltd., with a specification of 1 mL per vial and a viral titer of 3.0×10^10 PFU/mL.
  The investigational product is administered via two routes: intratumoral (IT) injection followed by intravenous (IV) infusion on Day 1 (D1) of each 21-day treatment cycle. Patients may receive up to 6 cycles of treatment.
  In this dose-escalation study, participants are enrolled into predefined dose cohorts. The starting dose for the first cohort is 6×10^10 PFU via intratumoral injection and 6×10^11 PFU via intravenous infusion.

SUMMARY:
This is a clinical study for patients with advanced solid tumors who have limited or no effective treatment options available. The study aims to evaluate a new investigational drug called VSV-02 Injection, which is developed by Shanghai Rongrui Pharmaceutical Technology Co., Ltd.

The main purpose of this open-label, single-arm study is to assess the preliminary effectiveness and safety of VSV-02 when it is given through two routes: directly into a vein (intravenously) and by injection directly into the tumor (intratumorally). Patients will receive the treatment on the first day of each 3-week cycle, for up to 6 cycles.

The study will follow a dose-escalation design to find a suitable dose. Treatment may be stopped if the disease progresses, if side effects become intolerable, or if the patient chooses to withdraw, among other reasons. Researchers will closely monitor patients to see if VSV-02 can help control the cancer and to record any side effects that may occur.

DETAILED DESCRIPTION:
1. Background Cancer remains a major public health concern worldwide. Despite advances in multimodal therapies including surgery, chemotherapy, radiotherapy, and targeted agents, effective treatments for recurrent or metastatic solid tumors are still limited. Immunotherapy, particularly immune checkpoint inhibitors (ICIs) targeting PD-1/PD-L1, has revolutionized oncology, but primary and acquired resistance remain significant challenges.

   Oncolytic viruses (OVs) represent a promising strategy to enhance antitumor immunity and overcome resistance. VSV-02 is an attenuated Vesicular Stomatitis Virus engineered to encode a CD3/PD-L1 bispecific antibody. It selectively infects and lyses tumor cells (oncolysis) and locally expresses the bispecific antibody, which bridges T cells and PD-L1-positive tumor cells to force T-cell activation and counteract PD-1/PD-L1-mediated suppression. This dual mechanism of action aims to stimulate a potent, localized immune response, making VSV-02 a compelling candidate for cancer immunotherapy.
2. Objectives Primary Objectives: To evaluate the preliminary efficacy of VSV-02 Injection administered via intravenous (IV) and intratumoral (IT) routes in subjects with advanced solid tumors, as measured by Objective Response Rate (ORR), Disease Control Rate (DCR), Duration of Response (DoR), Progression-Free Survival (PFS), and Overall Survival (OS) per RECIST 1.1.

   Secondary Objectives: To assess the safety and tolerability profile of VSV-02 (IV and IT), including the incidence and characteristics of adverse events (AEs), and changes in laboratory parameters, vital signs, ECGs, and physical examinations.
3. Study Design Trial Phase: Phase I Intervention Model: Single Group Assignment Allocation: Non-Randomized Masking: None (Open-Label) Primary Purpose: Treatment This is a single-arm, open-label, dose-escalation study. The study will follow a standard "3+3" design to evaluate the safety and preliminary efficacy of VSV-02.
4. Eligibility Criteria Age: ≥ 18 years. Diagnosis: Histologically or cytologically confirmed advanced solid tumors (e.g., melanoma, head and neck squamous cell carcinoma, cervical cancer, osteosarcoma, nasopharyngeal carcinoma, breast cancer, lung cancer, colorectal cancer, liver cancer, gastric cancer).

   Prior Therapy: Disease progression after at least two prior standard systemic therapies (including targeted therapy, where applicable), or for whom no standard therapy exists. Specific requirements vary by tumor type.

   Measurable Disease: At least one measurable lesion per RECIST 1.1 and at least one lesion accessible for IT injection.

   Performance Status: ECOG score of 0-2 and life expectancy ≥ 12 weeks. Organ Function: Adequate hematological, hepatic, and renal function. Key exclusion criteria include: symptomatic or untreated brain metastases (asymptomatic, stable for ≥3 months post-treatment allowed); active autoimmune disease; significant cardiovascular disease; active infection; concurrent anticoagulant therapy; and requirement for high-dose systemic corticosteroids.
5. Interventions Participants will receive VSV-02 Injection (supplied by Shanghai Rongrui Pharmaceutical Technology Co., Ltd.; specification: 1mL/vial; titer: 3.0×10^10 PFU/mL) on Day 1 of each 21-day cycle for up to 6 cycles. Dosing involves concurrent IV and IT administration. The starting dose level is 6×10^10 PFU (IT) + 6×10^11 PFU (IV). The IT injection volume will be determined based on tumor size measured within 24 hours prior to injection, with a maximum total volume of 10 mL per subject per day. Treatment continues until disease progression (with clinical deterioration), unacceptable toxicity, withdrawal of consent, completion of 6 cycles, or other protocol-specified criteria.
6. Outcome Measures Efficacy Assessments: Tumor assessments will be performed per RECIST 1.1. Subjects with initial radiographic progression per RECIST 1.1 but without clinical deterioration may continue treatment, with progression confirmed per iRECIST ≥4 weeks later. Primary efficacy endpoints are ORR, DCR, DoR, PFS, and OS.

Safety Assessments: Safety will be monitored throughout the study. AEs will be graded according to NCI CTCAE v5.0. Assessments include monitoring of AEs/SAEs, DLTs/MTD, clinical laboratory tests, vital signs, ECGs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

Voluntary signed informed consent.

Age ≥ 18 years.

Histologically or cytologically confirmed advanced solid tumor (e.g., melanoma, head and neck squamous cell carcinoma, cervical cancer, osteosarcoma, nasopharyngeal carcinoma, breast cancer, lung cancer, colorectal cancer, liver cancer, gastric cancer).

Disease progression after at least two prior lines of standard therapy (including targeted therapy), or for whom no standard therapy exists or is medically unsuitable.

At least one measurable lesion per RECIST 1.1 criteria.

At least one lesion accessible for intratumoral injection.

ECOG performance status of 0-2.

Life expectancy ≥ 12 weeks.

Adequate organ and bone marrow function.

Negative pregnancy test for women of childbearing potential.

Agreement to use effective contraception during the study and for at least 6 months after the last dose.

Exclusion Criteria:

Symptomatic or untreated brain metastases (asymptomatic or stable for ≥3 months after local therapy allowed).

Radiotherapy to the target lesion within 2 months.

History of other active malignancy within 5 years (with specific exceptions).

Lesion intended for injection with a longest diameter > 100 mm.

Participation in another interventional clinical trial within 4 weeks.

Prior or planned organ/tissue transplantation.

Active HIV, Hepatitis B, Hepatitis C, or Syphilis infection meeting specific criteria.

Requirement for concomitant antiviral or therapeutic anticoagulation.

Uncontrolled ≥ Grade 3 active infection.

Specific washout periods for prior anti-cancer therapies not met.

Uncontrolled cardiovascular disease.

Active or history of autoimmune disease (with specific exceptions).

Requirement for systemic corticosteroids (>10 mg prednisone equivalent) within 14 days or during the study.

Tumors located in high-risk anatomical sites.

Administration of live vaccines during the study period.

Known hypersensitivity to any component of the study drug or related immunotherapies.

History of severe mental illness, substance abuse, or other conditions that may interfere with study compliance.

Pregnancy or lactation.

Toxicities from previous anti-cancer therapy not recovered to ≤ Grade 1 (except alopecia).

Any other condition deemed inappropriate for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment until the first occurrence of disease progression or the end of treatment, up to 24 months.
  ORR is defined as the proportion of participants achieving a best overall response of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as assessed by the investigator.
Disease Control Rate (DCR) | From enrollment until the first occurrence of disease progression or the end of treatment, up to 24 months.
  DCR is defined as the proportion of participants achieving a best overall response of complete response (CR), partial response (PR), or stable disease (SD) (lasting for at least 6 weeks) per RECIST 1.1.
Duration of Response (DoR) | From the first objective response (CR or PR) until disease progression or death from any cause, assessed up to 36 months.
  DoR is defined as the time from the first documentation of CR or PR to the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first, as per RECIST 1.1.
Progression-Free Survival (PFS) | From enrollment until the first occurrence of disease progression or death from any cause, assessed up to 36 months.
  PFS is defined as the time from enrollment to the first documentation of progressive disease (PD) as per RECIST 1.1 or death from any cause, whichever occurs first.
verall Survival (OS) | From enrollment until death from any cause, assessed up to 60 months.
  OS is defined as the time from enrollment to death due to any cause.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | From first dose of study drug until 30 days after the last dose, up to 7 months.
  The incidence and severity of AEs will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: LiuZhong Yang, master, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT07260591/Prot_SAP_000.pdf